CLINICAL TRIAL: NCT05164198
Title: Multicenter, Prospective Clinical Trial for Optimizing TNF Inhibitor Dose Adjustment in Ankylosing Spondylitis Patients With Stable Disease Activity
Brief Title: REduCed Dose of TNFi in Patients With Ankylosing SpondyliTis (RECAST)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hanyang University Seoul Hospital (Other)
Collaborators: Linical Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HC21C0076
Record Dates: First submitted 2021-11-08; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-10

CONDITIONS: Ankylosing Spondylitis; Axial Spondyloarthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Axial Spondyloarthritis | interventions — Adalimumab; Etanercept; golimumab; CT-P13

STUDY DESIGN:
Intervention Model Description: Phase 4, randomized, parallel, non-inferiority, open-label, multi-center clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open-label reduced-dose TNFi (Experimental): Participants in the experimental arm will receive one of the intervention below according to the TNFi agent used at baseline:
  1. Adalimumab 40mg subcutaneous every 3 weeks (Q3W) from week 0 to week 48.
  2. Etanercept 50mg subcutaneous every 10 days (Q10D) from week 0 to week 48.
  3. Golimumab 50mg (100mg if a participant's body weight ≥ 100kg) subcutaneous every 5 weeks (Q5W) from week 0 to week 48.
  4. Remsima SC 120mg subcutaneous every 3 weeks (Q3W) from week 0 to week 48.
  Interventions: Biological: Adalimumab and its biosimilars; Biological: Biological: Etanercept and its biosimilars; Biological: Golimumab; Biological: Infliximab biosimilar
- Open-label full-dose TNFi (Active Comparator): Participants in the comparator arm will receive one of the intervention below according to the TNFi agent used at baseline:
  1. Adalimumab 40mg subcutaneous every 2 weeks (Q2W) from week 0 to week 48.
  2. Etanercept 50mg subcutaneous every week (QW) from week 0 to week 48.
  3. Golimumab 50mg (100mg if a participant's body weight ≥ 100kg) subcutaneous every 4 weeks (Q4W) from week 0 to week 48.
  4. Remsima SC 120mg subcutaneous every 2 weeks (Q2W) from week 0 to week 48.
  Interventions: Biological: Adalimumab and its biosimilars; Biological: Biological: Etanercept and its biosimilars; Biological: Golimumab; Biological: Infliximab biosimilar

INTERVENTIONS:
Biological: Adalimumab and its biosimilars — 1. Active substance: Adalimumab
  2. Pharmaceutical form: Prefilled syringe
  3. Concentration: 100mg/mL
  4. Route of administration: Subcutaneous injection
  Other Names: Humira; Adaloce
Biological: Biological: Etanercept and its biosimilars — 1. Active substance: Etanercept
  2. Pharmaceutical form: Prefilled syringe
  3. Concentration: 50mg/mL
  4. Route of administration: Subcutaneous injection
  Other Names: Enbrel; Eucept; Etalace
Biological: Golimumab — 1. Active substance: Adalimumab
  2. Pharmaceutical form: Prefilled syringe
  3. Concentration: 100mg/mL
  4. Route of administration: Subcutaneous injection
  Other Names: Simponi
Biological: Infliximab biosimilar — 1. Active substance: Infliximab
  2. Pharmaceutical form: Prefilled syringe
  3. Concentration: 120mg/mL
  4. Route of administration: Subcutaneous injection
  Other Names: Remsima

SUMMARY:
Participants maintaining stable disease activity of Ankylosing Spondylitis (AS) with standard-dose tumor necrosis factor inhibitor (TNFi) treatment will randomly split into two groups: maintaining standard-dose TNFi, versus reduced-dose TNFi. The proportion of participants not underwent flare between the two groups will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Ankylosing spondylitis (AS) and meet the modified New York classification criteria for AS.
* Subjects maintaining stable disease (Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] < 4) with standard-dose subcutaneous tumor-necrosis factor inhibitor (TNFi) treatment during previous 6 months from screening.
* Ankylosing Spondylitis Disease Activity Score (ASDAS) < 2.1 at screening and 12 weeks prior to screening
* In subjects treated with methotrexate or sulfasalazine, the dose should be maintained (methotrexate≤ 25mg/day, sulfasalazine ≤ 3 g/day) during previous 4 weeks before screening.
* In subjects treated with systemic glucocorticoids, the dose should be less than 10mg/day of predinisolone or equivalent during at least 2 weeks from the screening
* Subjects with stable dose of concomitant NSAID (including Cox2 inhibitors) during the 2 weeks from the randomization

Exclusion Criteria:

* Exposure to more than 1 TNFi
* History of hypersensitivity reaction to any TNFis
* Subjects with concomitant fibromyalgia, as determined by the investigator
* Subjects who have received any TNFis with reduced dosage
* Presence of total spinal ankylosis ('Bamboo spine')
* Female subjects who are breastfeeding, pregnant, or plan to become pregnant during the study
* Subjects with a history of malignancies and lymphoproliferative disorder including lymphoma within 5 years (Basal cell carcinoma treated within previous 3 months and showing no evidence of recurrence, actinic keratosis, and treated cervical/colon carcinoma in situ were allowed.)
* Subjects with current or history of severe, progressive, and/or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac or neurological disease, as determined by the investigator
* Subjects with significant laboratory abnormalities included but not limited to:

  1. AST/ALT > 3.0 X ULN
  2. White blood cell (WBC) < 3000/μL and/or absolute neutrophil count (ANC) < 1500/μL
  3. Platelet count <100,000/μL and/or hemoglobin level <8.5 g/dL
  4. Serum creatinine ≥ 1.5 X ULN
* Subjected with any high-potency opioids (ex. methadone, hydromorphone, morphine, oxycodone, oxymorphone, fentanyl, levorphanol, buprenorphine, meperidine)
* Subjects with current acute or chronic viral hepatitis B or C or with human immunodeficiency virus (HIV) infection
* Subjects planning to receive any live attenuated vaccinations after screening
* Subjects has history of chronic alcohol abuse or drug abuse within 6 months from screening
* Subjects concomitantly treated with systemic glucocorticoid (>10mg/day of prednisolone or equivalent doses)
* Subjects with any other condition that, in the Investigator's judgment, would make the subject unsuitable for inclusion in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Estimated)
Dates: Start 2022-01-15 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who did not experience a flare | From week 0 to week 48
  Flare is defined as below:
  * A participant was considered to have experienced a flare if the participant had an Ankylosing spondylitis disease activity score (ASDAS) greater or equal to (≥ 2.1) at 2 consecutive visits or an ASDAS greater than (> 3.5) at any visit.
  * If a participant had an ASDAS ≥ 2.1 and ≤ 3.5, the participant has an additional visit 4 weeks later and ASDAS is assessed by the investigator to confirm the flare.
  The ASDAS was calculated as the sum of the following components: 0.121 x Back pain (BASDAI Q2 result) 0.058 x Duration of morning stiffness (BASDAI Q6 result) 0.110 x PGADA (Patient's Global Assessment of Disease Activity) 0.073 x Peripheral pain/swelling (BASDAI Q3 result) 0.579 × (natural logarithm [ln] of the (CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue were all assessed on a numerical scale (0 to 10 units). Higher scores mean a worse outcome in the all following components.

SECONDARY OUTCOMES:
Change from baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at week 12. | Week 12
  The ASDAS was calculated as the sum of the following components: 0.121 x Back pain (BASDAI Q2 result) 0.058 x Duration of morning stiffness (BASDAI Q6 result) 0.110 x PGADA (Patient's Global Assessment of Disease Activity) 0.073 x Peripheral pain/swelling (BASDAI Q3 result) 0.579 × (natural logarithm [ln] of the (CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue were all assessed on a numerical scale (0 to 10 units). Higher scores mean a worse outcome in the all following components.
Change from baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at week 24. | Week 24
  The ASDAS was calculated as the sum of the following components: 0.121 x Back pain (BASDAI Q2 result) 0.058 x Duration of morning stiffness (BASDAI Q6 result) 0.110 x PGADA (Patient's Global Assessment of Disease Activity) 0.073 x Peripheral pain/swelling (BASDAI Q3 result) 0.579 × (natural logarithm [ln] of the (CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue were all assessed on a numerical scale (0 to 10 units). Higher scores mean a worse outcome in the all following components.
Change from baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at week 36. | Week 36
  The ASDAS was calculated as the sum of the following components: 0.121 x Back pain (BASDAI Q2 result) 0.058 x Duration of morning stiffness (BASDAI Q6 result) 0.110 x PGADA (Patient's Global Assessment of Disease Activity) 0.073 x Peripheral pain/swelling (BASDAI Q3 result) 0.579 × (natural logarithm [ln] of the (CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue were all assessed on a numerical scale (0 to 10 units). Higher scores mean a worse outcome in the all following components.
Change from baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at week 48. | Week 48
  The ASDAS was calculated as the sum of the following components: 0.121 x Back pain (BASDAI Q2 result) 0.058 x Duration of morning stiffness (BASDAI Q6 result) 0.110 x PGADA (Patient's Global Assessment of Disease Activity) 0.073 x Peripheral pain/swelling (BASDAI Q3 result) 0.579 × (natural logarithm [ln] of the (CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue were all assessed on a numerical scale (0 to 10 units). Higher scores mean a worse outcome in the all following components.
Change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at week 12. | Week 12
  The BASDAI is a validated self-reported instrument, which consists of six 10 unit horizontal Numeric Rating Scales (NRS) to measure the disease activity of ankylosing spondylitis (AS) from the subject's perspective. It measures the severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration) over the last week. The final BASDAI scores ranges from 0 to 10, with lower scores indicating lower disease activity.
Change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at week 24. | Week 24
  The BASDAI is a validated self-reported instrument, which consists of six 10 unit horizontal Numeric Rating Scales (NRS) to measure the disease activity of ankylosing spondylitis (AS) from the subject's perspective. It measures the severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration) over the last week. The final BASDAI scores ranges from 0 to 10, with lower scores indicating lower disease activity.
Change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at week 36. | Week 36
  The BASDAI is a validated self-reported instrument, which consists of six 10 unit horizontal Numeric Rating Scales (NRS) to measure the disease activity of ankylosing spondylitis (AS) from the subject's perspective. It measures the severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration) over the last week. The final BASDAI scores ranges from 0 to 10, with lower scores indicating lower disease activity.
Change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at week 48. | Week 48
  The BASDAI is a validated self-reported instrument, which consists of six 10 unit horizontal Numeric Rating Scales (NRS) to measure the disease activity of ankylosing spondylitis (AS) from the subject's perspective. It measures the severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration) over the last week. The final BASDAI scores ranges from 0 to 10, with lower scores indicating lower disease activity.
Percentage of participants with Axial SpondyloArthritis International Society 20 % Response Criteria (ASAS20) Response at week 12. | Week 12
  The ASAS20 response was defined as an improvement of at least 20 % and absolute improvement of at least 1 unit on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and absence of deterioration in the potential remaining domain [deterioration was defined as a relative worsening of at least 20 % and an absolute worsening of at least 1 unit]. Higher scores mean a worse outcome in the all domains.
Percentage of participants with Axial SpondyloArthritis International Society 20 % Response Criteria (ASAS20) Response at week 24. | Week 24
  The ASAS20 response was defined as an improvement of at least 20 % and absolute improvement of at least 1 unit on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and absence of deterioration in the potential remaining domain [deterioration was defined as a relative worsening of at least 20 % and an absolute worsening of at least 1 unit]. Higher scores mean a worse outcome in the all domains.
Percentage of participants with Axial SpondyloArthritis International Society 20 % Response Criteria (ASAS20) Response at week 36. | Week 36
  The ASAS20 response was defined as an improvement of at least 20 % and absolute improvement of at least 1 unit on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and absence of deterioration in the potential remaining domain [deterioration was defined as a relative worsening of at least 20 % and an absolute worsening of at least 1 unit]. Higher scores mean a worse outcome in the all domains.
Percentage of participants with Axial SpondyloArthritis International Society 20 % Response Criteria (ASAS20) Response at week 48. | Week 48
  The ASAS20 response was defined as an improvement of at least 20 % and absolute improvement of at least 1 unit on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and absence of deterioration in the potential remaining domain [deterioration was defined as a relative worsening of at least 20 % and an absolute worsening of at least 1 unit]. Higher scores mean a worse outcome in the all domains.
Percentage of participants with Axial SpondyloArthritis International Society 40 % Response Criteria (ASAS40) Response at week 12. | Week 12
  The ASAS40 response was defined as a relative improvement of at least 40 % and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and no worsening at all in the remaining domain. Higher scores mean a worse outcome in the all domains.
Percentage of participants with Axial SpondyloArthritis International Society 40 % Response Criteria (ASAS40) Response at week 24. | Week 24
  The ASAS40 response was defined as a relative improvement of at least 40 % and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and no worsening at all in the remaining domain. Higher scores mean a worse outcome in the all domains.
Percentage of participants with Axial SpondyloArthritis International Society 40 % Response Criteria (ASAS40) Response at week 36. | Week 36
  The ASAS40 response was defined as a relative improvement of at least 40 % and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and no worsening at all in the remaining domain. Higher scores mean a worse outcome in the all domains.
Percentage of participants with Axial SpondyloArthritis International Society 40 % Response Criteria (ASAS40) Response at week 48. | Week 48
  The ASAS40 response was defined as a relative improvement of at least 40 % and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and no worsening at all in the remaining domain. Higher scores mean a worse outcome in the all domains.
Percentage of participants with Axial SpondyloArthritis International Society 5/6 Response Criteria (ASAS5/6) Response at week 12. | Week 12
  The ASAS 5/6 response was defined as achieving at least 20 % improvement in 5 of 6 domains, including the 4 domains defined for ASAS20 as well as spinal mobility (lateral spinal flexion) and C-reactive Protein (CRP).
Percentage of participants with Axial SpondyloArthritis International Society 5/6 Response Criteria (ASAS5/6) Response at week 24. | Week 24
  The ASAS 5/6 response was defined as achieving at least 20 % improvement in 5 of 6 domains, including the 4 domains defined for ASAS20 as well as spinal mobility (lateral spinal flexion) and C-reactive Protein (CRP).
Percentage of participants with Axial SpondyloArthritis International Society 5/6 Response Criteria (ASAS5/6) Response at week 36. | Week 36
  The ASAS 5/6 response was defined as achieving at least 20 % improvement in 5 of 6 domains, including the 4 domains defined for ASAS20 as well as spinal mobility (lateral spinal flexion) and C-reactive Protein (CRP).
Percentage of participants with Axial SpondyloArthritis International Society 5/6 Response Criteria (ASAS5/6) Response at week 48. | Week 48
  The ASAS 5/6 response was defined as achieving at least 20 % improvement in 5 of 6 domains, including the 4 domains defined for ASAS20 as well as spinal mobility (lateral spinal flexion) and C-reactive Protein (CRP).
Percentage of participants with Axial SpondyloArthritis International Society Partial Remission Response Criteria (ASAS-PR) Response at week 12. | Week 12
  The ASAS partial remission (PR) response was defined as a score of ≤ 2 units on a 0 to 10 unit scale in all 4 domains listed for ASAS20.
Percentage of participants with Axial SpondyloArthritis International Society Partial Remission Response Criteria (ASAS-PR) Response at week 24. | Week 24
  The ASAS partial remission (PR) response was defined as a score of ≤ 2 units on a 0 to 10 unit scale in all 4 domains listed for ASAS20.
Percentage of participants with Axial SpondyloArthritis International Society Partial Remission Response Criteria (ASAS-PR) Response at week 36. | Week 36
  The ASAS partial remission (PR) response was defined as a score of ≤ 2 units on a 0 to 10 unit scale in all 4 domains listed for ASAS20.
Percentage of participants with Axial SpondyloArthritis International Society Partial Remission Response Criteria (ASAS-PR) Response at week 48. | Week 48
  The ASAS partial remission (PR) response was defined as a score of ≤ 2 units on a 0 to 10 unit scale in all 4 domains listed for ASAS20.
Change from baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at week 12. | Week 12
  The BASFI is a validated disease-specific instrument for assessing physical function. The BASFI comprises 10 items relating to the past week. The BASFI is the mean of the 10 scores such that the total score ranges from 0 (Easy) to 10 (Impossible), with lower scores indicating better physical function. The change from Week 0 is calculated, a negative value indicating improvement and a positive value worsening.
Change from baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at week 24. | Week 24
  The BASFI is a validated disease-specific instrument for assessing physical function. The BASFI comprises 10 items relating to the past week. The BASFI is the mean of the 10 scores such that the total score ranges from 0 (Easy) to 10 (Impossible), with lower scores indicating better physical function. The change from Week 0 is calculated, a negative value indicating improvement and a positive value worsening.
Change from baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at week 36. | Week 36
  The BASFI is a validated disease-specific instrument for assessing physical function. The BASFI comprises 10 items relating to the past week. The BASFI is the mean of the 10 scores such that the total score ranges from 0 (Easy) to 10 (Impossible), with lower scores indicating better physical function. The change from Week 0 is calculated, a negative value indicating improvement and a positive value worsening.
Change from baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at week 48. | Week 48
  The BASFI is a validated disease-specific instrument for assessing physical function. The BASFI comprises 10 items relating to the past week. The BASFI is the mean of the 10 scores such that the total score ranges from 0 (Easy) to 10 (Impossible), with lower scores indicating better physical function. The change from Week 0 is calculated, a negative value indicating improvement and a positive value worsening.
Change from baseline in Bath Ankylosing Spondylitis Disease Metrology Index (BASMI) at week 24. | Week 24
  The BASMI is a disease-specific measure consisting of 5 clinical measures to reflect subject axial status: cervical rotation; tragus to wall distance; lateral lumbar flexion; lumbar flexion (modified Schober test); intermalleolar distance. According to the linear definition of the BASMI a score of 0 to 10 was calculated for each item based on the measurement. The mean of the sum of the 5 scores provided the total BASMI score, ranging from 0 to 10. The higher the BASMI score the more severe the patient's limitation of movement due to their axial spondyloarthritis (axSpA). The change from Week 0 is calculated, a negative value indicating improvement and a positive value worsening.
Change from baseline in Bath Ankylosing Spondylitis Disease Metrology Index (BASMI) at week 48. | Week 48
  The BASMI is a disease-specific measure consisting of 5 clinical measures to reflect subject axial status: cervical rotation; tragus to wall distance; lateral lumbar flexion; lumbar flexion (modified Schober test); intermalleolar distance. According to the linear definition of the BASMI a score of 0 to 10 was calculated for each item based on the measurement. The mean of the sum of the 5 scores provided the total BASMI score, ranging from 0 to 10. The higher the BASMI score the more severe the patient's limitation of movement due to their axial spondyloarthritis (axSpA). The change from Week 0 is calculated, a negative value indicating improvement and a positive value worsening.
Change from baseline in Masstricht Ankylosing Spondylitis Enthesitis Score (MASES) at week 24. | Week 24
  The Masstricht Ankylosing Spondylitis Enthesitis Score (MASES) is a disease-specific measure to assess the level of enthesitis in Ankylosing Spondylitis. It is based on clinical examination by assessor who determined by presence (score 1) or absence (score 0) of enthesitis at 13 different sites as below:
  * Both 1st costochondral
  * Both 7th costochondral
  * Both iliac crest
  * Both anterior superior iliac spine
  * Both posterior superior iliac spine
  * Both proximal Achilles tendon
  * 5th lumbar spinous process
Change from baseline in Masstricht Ankylosing Spondylitis Enthesitis Score (MASES) at week 48. | Week 48
  The Masstricht Ankylosing Spondylitis Enthesitis Score (MASES) is a disease-specific measure to assess the level of enthesitis in Ankylosing Spondylitis. It is based on clinical examination by assessor who determined by presence (score 1) or absence (score 0) of enthesitis at 13 different sites as below:
  * Both 1st costochondral
  * Both 7th costochondral
  * Both iliac crest
  * Both anterior superior iliac spine
  * Both posterior superior iliac spine
  * Both proximal Achilles tendon
  * 5th lumbar spinous process
Change from baseline in swollen/tender joint count (0-44) at week 24. | Week 24
  American College of Rheumatology (ACR), swollen joint count were an assessment of 44 joints. Joints are classified as either swollen or not swollen (tender or non-tender). An increase in swollen joints from baseline represented disease progression and/or joint worsening.
Change from baseline in swollen/tender joint count (0-44) at week 48. | Week 48
  American College of Rheumatology (ACR), swollen joint count were an assessment of 44 joints. Joints are classified as either swollen or not swollen (tender or non-tender). An increase in swollen joints from baseline represented disease progression and/or joint worsening.
Change from baseline in Erythrocyte sedimentation rate (ESR) at week 12. | Week 12
Change from baseline in Erythrocyte sedimentation rate (ESR) at week 24. | Week 24
Change from baseline in Erythrocyte sedimentation rate (ESR) at week 36. | Week 36
Change from baseline in Erythrocyte sedimentation rate (ESR) at week 48. | Week 48
Change from baseline in serum C-Reactive Protein (CRP) level at week 12. | Week 12
Change from baseline in serum C-Reactive Protein (CRP) level at week 24. | Week 24
Change from baseline in serum C-Reactive Protein (CRP) level at week 36. | Week 36
Change from baseline in serum C-Reactive Protein (CRP) level at week 48. | Week 48
Change from baseline in Assessment of SpondyloArthritis international Society (ASAS)-health index (ASAS-HI) at week 24. | Week 24
  The self-report questionnaire measures functioning and health across 17 aspects of health and 9 environmental factors (EF) in patients with spondyloarthritis. The ASAS HI contains items addressing categories of pain, emotional functions, sleep, sexual function, mobility, self care, and community life.
Change from baseline in Assessment of SpondyloArthritis international Society (ASAS)-health index (ASAS-HI) at week 48. | Week 48
  The self-report questionnaire measures functioning and health across 17 aspects of health and 9 environmental factors (EF) in patients with spondyloarthritis. The ASAS HI contains items addressing categories of pain, emotional functions, sleep, sexual function, mobility, self care, and community life.
Change from baseline in 5-level EQ-5D version (EQ-5D-5L) at week 24. | Week 24
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Change from baseline in 5-level EQ-5D version (EQ-5D-5L) at week 48. | Week 48
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
The amount of NSAID intake between week 0 and 12 | From week 0 to week 12
  The general formula for the calculation is:
  (equivalent NSAID score) × (days of intake during period of interest) × (days with intake per week)/(period of interest in days)
  1. Equivalent NSAID score 0 = no intake 100 = 150mg diclofenac / 1000mg naproxen / 200mg aceclofenac / 400mg celecoxib / 600mg etodolac / 150mg indomethacin / 15mg meloxicam / 20mg piroxicam
  2. A scale indicating days with intake per week 0 = did not take any NSAID in a week 0.5/7 = ≤1 day in a week 2/7 = >1 and ≤3 days in a week 4/7 = >3 and ≤5 days in a week 6/7 = >5 days in a week 1 = every day
  3. days of intake during the period of interest
  For example, if during a period of interest of 12 weeks, the patient has taken piroxicam 20 mg for 8 weeks and if during this 8-week period he has taken piroxicam 3-5 days per week the calculation is as follows:
  100 (20 mg piroxicam score) × 56 (8 weeks) × 4/7 (3-5 days/week)/84 (12 weeks) = 38.1
The amount of NSAID intake between week 12 and 24 | From week 12 to week 24
  The general formula for the calculation is:
  (equivalent NSAID score) × (days of intake during period of interest) × (days with intake per week)/(period of interest in days)
  1. Equivalent NSAID score 0 = no intake 100 = 150mg diclofenac / 1000mg naproxen / 200mg aceclofenac / 400mg celecoxib / 600mg etodolac / 150mg indomethacin / 15mg meloxicam / 20mg piroxicam
  2. A scale indicating days with intake per week 0 = did not take any NSAID in a week 0.5/7 = ≤1 day in a week 2/7 = >1 and ≤3 days in a week 4/7 = >3 and ≤5 days in a week 6/7 = >5 days in a week 1 = every day
  3. days of intake during the period of interest
  For example, if during a period of interest of 12 weeks, the patient has taken piroxicam 20 mg for 8 weeks and if during this 8-week period he has taken piroxicam 3-5 days per week the calculation is as follows:
  100 (20 mg piroxicam score) × 56 (8 weeks) × 4/7 (3-5 days/week)/84 (12 weeks) = 38.1
The amount of NSAID intake between week 24 and 36 | From week 24 to week 36
  The general formula for the calculation is:
  (equivalent NSAID score) × (days of intake during period of interest) × (days with intake per week)/(period of interest in days)
  1. Equivalent NSAID score 0 = no intake 100 = 150mg diclofenac / 1000mg naproxen / 200mg aceclofenac / 400mg celecoxib / 600mg etodolac / 150mg indomethacin / 15mg meloxicam / 20mg piroxicam
  2. A scale indicating days with intake per week 0 = did not take any NSAID in a week 0.5/7 = ≤1 day in a week 2/7 = >1 and ≤3 days in a week 4/7 = >3 and ≤5 days in a week 6/7 = >5 days in a week 1 = every day
  3. days of intake during the period of interest
  For example, if during a period of interest of 12 weeks, the patient has taken piroxicam 20 mg for 8 weeks and if during this 8-week period he has taken piroxicam 3-5 days per week the calculation is as follows:
  100 (20 mg piroxicam score) × 56 (8 weeks) × 4/7 (3-5 days/week)/84 (12 weeks) = 38.1
The amount of NSAID intake between week 36 and 48 | From week 36 to week 48
  The general formula for the calculation is:
  (equivalent NSAID score) × (days of intake during period of interest) × (days with intake per week)/(period of interest in days)
  1. Equivalent NSAID score 0 = no intake 100 = 150mg diclofenac / 1000mg naproxen / 200mg aceclofenac / 400mg celecoxib / 600mg etodolac / 150mg indomethacin / 15mg meloxicam / 20mg piroxicam
  2. A scale indicating days with intake per week 0 = did not take any NSAID in a week 0.5/7 = ≤1 day in a week 2/7 = >1 and ≤3 days in a week 4/7 = >3 and ≤5 days in a week 6/7 = >5 days in a week 1 = every day
  3. days of intake during the period of interest
  For example, if during a period of interest of 12 weeks, the patient has taken piroxicam 20 mg for 8 weeks and if during this 8-week period he has taken piroxicam 3-5 days per week the calculation is as follows:
  100 (20 mg piroxicam score) × 56 (8 weeks) × 4/7 (3-5 days/week)/84 (12 weeks) = 38.1
Percentage of patients at Least One Adverse Event (AE) During the study period. | From week 0 and week 48
  An AE was any untoward medical occurrence in a patient or clinical investigation study participant administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Hwan Kim, MD, PhD, Principal Investigator — Hanyang University